CLINICAL TRIAL: NCT05063084
Title: A Randomised Controlled Trial Comparing Pre-oxygenation Strategies With High-flow Humidified Nasal Oxygenation Versus Apnoeic Facemask Oxygenation During Rapid Sequence Induction in Children Aged Less Then 11 Years
Brief Title: High-flow Nasal Cannula Oxygenation During Rapid Sequence Induction in Children
Acronym: OPTINECK
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP201164; 2021-A01419-32 (Other: ID-RCB Number)
Record Dates: First submitted 2021-08-04; First posted 2021-09-30 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Pediatric Surgery; Rapid Sequence Induction
Keywords: nasal high flow oxygen; rapid sequence induction; preoxygenation; pediatric
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OHD (HFNO) (Experimental): High flow nasal oxygen
  Interventions: Procedure: Optiflow - HFNO
- Control (Other): Classic pre-oxygenation with facemask
  Interventions: Procedure: Classic

INTERVENTIONS:
Procedure: Optiflow - HFNO — Pre-oxygenation: HFNO with a 2 L/Kg/min flow during 2 min with 100% FiO2 Oxygenation: during the tracheal intubation, HFNO with a 2 L/Kg/min flow during 2 min with 100% FiO2
  Other Names: OHD (Oxygenation Haut Débit)
  Arms: OHD (HFNO)
Procedure: Classic — Pre-oxygenation: with facemask during 2 min with 100% FiO2, flow 6 to 8L/min. No oxygenation during the tracheal intubation
  Arms: Control

SUMMARY:
This randomised study aims to compare the utilization of high-flow humidified nasal oxygenation (HFNO) with standard care, using apnoeic facemask oxygenation, during rapid sequence induction (RSI) of anesthesia in young children.

170 children aged less then 11 years, admitted to the operating room for surgery and with a medical indication of a RSI of anesthesia will be recruited in one university hospital (Necker-Enfants-Malades in Paris).

Children will be randomly assigned into two groups: the control group will benefit of standard care and the HFNO group will receive heated and humidified oxygen through a nasal cannula device during pre-oxygenation and apnoea time prior to tracheal intubation.

HFNO has been evaluated and showed benefits in rapid sequence induction of anesthesia in adults and prolonged apnea time before desaturation in children. To the investigators' knowledge the potential benefit of HFNO during RSI in young children remain to be evaluated.

DETAILED DESCRIPTION:
Hypoxic events during rapid sequence induction (RSI) in children remain more frequent than during standard induction. Although the exact incidence is difficult to appreciate. However the deleterious consequences of hypoxemia during tracheal intubation procedures are well known.

HFNO is an effective technique to supplement oxygen including during apnoea. Studies in children have shown benefits both during breathing and apneic situation.

A monocentric controlled randomized study including children, aged less then 11 years, will be conducted in order to assess the potential benefits of this technique during RSI. The rate of successful tracheal intubation without oxygen desaturation is the primary outcome.

Children will be randomly assigned into two groups:

* The control group will benefit of standard RSI. Pre-oxygenation will be given through facemask with 100% oxygen during 2 minutes, with a flow of 6 to 8 L.min-1 depending on the age of the child. No oxygen will be delivered during laryngoscopy.
* The HFNO group will be given 2 L.Kg-1.min-1 of humidified and heated 100% O2 through a nasal cannula during a 2 minutes pre-oxygenation and then throughout laryngoscopy.

Adverse events will be recorded and follow-up continued until discharge from the post anesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* child from birth until 10 years
* patient needing (elective or in emergency) surgery under general anesthesia requiring tracheal intubation and fulfilling all criteria for a rapid sequence induction
* Parents or legal guardians signed the Informed consent form
* Social insurance affiliation

Exclusion Criteria

- child having one or more contraindication to use high flow nasal oxygenation:

* Nasal obstruction
* Recent trauma of aero-digestives tracts
* Epistaxis
* Known or suspected fracture of the skull base
* Cephalo-spinal fluid leak or all other communication between nasal space and intracranial space
* Tuberculosis or other nasal or lung infection
* Pneumothorax or pneumo-mediastin documented or suspected
* Complete limitation of mouth opening

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Intubation without oxygen desaturation episode | Up to 10 minutes
  Intubation without oxygen desaturation episode, defined as pulsed oxymetry <95% during the rapid sequence induction process of anesthesia in the operating room.

SECONDARY OUTCOMES:
Oxygen saturation level | Up to 10 minutes
  Measurement of the lowest oxygen saturation during the tracheal intubation process
Tracheal intubation without facemask reventilation | Up to 10 minutes
  Tracheal intubation without facemask reventilation
Number of attempted tracheal intubations required to succeed the process | Up to 10 minutes
  Number of attempted tracheal intubations required to succeed the process
Occurrence of all adverse events | until the exit of the recovery room
  Occurrence of all adverse events during tracheal intubation in the operating room (linked or not to the use of HFNO)
Satisfaction of the anaesthetist and the anaesthesia team regarding the use of HFNO | Exit of the recovery room
  Questionnaire about satisfaction, the use of the procedure, stress level and potential genes

CONTACTS AND LOCATIONS:
Overall Officials: Gilles ORLIAGUET, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker - Enfants malades, Paris, France

IPD SHARING:
Plan to Share IPD: No